CLINICAL TRIAL: NCT03517553
Title: Effects of Exercise Using Electrical Muscle Stimulation in End Stage Kidney Disease
Brief Title: Effects of Exercise by Neuromuscular Stimulation in Dialysis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study subjects that were enrolled all completed all visits. PI is currently unable to work on analyzing results
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201301731
Record Dates: First submitted 2017-02-19; First posted 2018-05-07 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Dialysis
Keywords: electrical muscle stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EMS users in ESRD (Experimental): Subjects then initiate passive electrical muscle stimulation (EMS) delivered by a commercially available FDA approved neuromuscular stimulator (EMPI 300PV or its replacement, EMPI Continuum device obtained from EMPI, Inc., St Paul MN) 3 times a week to the quadriceps muscle groups (15 minutes on each side, 30 minutes total) while on hemodialysis. The duration of training will last for 4 months. Subjects will be monitored at regular intervals during the training to make sure they are doing the training correctly and they are not experiencing any problems.
  Interventions: Device: EMS users in ESRD

INTERVENTIONS:
Device: EMS users in ESRD — use of passive electrical muscle stimulation on quadriceps muscle 3 times a week for patients in dialysis

SUMMARY:
The investigators propose a pilot feasibility study to determine if exercise delivered by passive electrical muscle stimulation (EMS) in patients with end stage renal disease (ESRD) on hemodialysis improves physical fitness and insulin resistance, outcome markers associated with morbidity and mortality in this population.

DETAILED DESCRIPTION:
Subjects who enroll and meet the inclusion and none of the exclusion criteria will first undergo baseline testing including recording of demographic, medical, dialysis and exercise history, taking surveys to assess quality of life and overall mood, measurement of vital signs and anthropomorphic measurements (height, weight, thigh circumference), have blood collected to assess insulin resistance and cytokine levels, measurement of distance walked in 6 minutes and testing of thigh muscle strength.

Subjects will then undergo a 1 month observation period to monitor and optimize their dialysis treatment.

After 1 month the subjects will undergo a repeat assessment of all the baseline testing. They will also undergo a standardized exercise stress test and measurement of body fat and lean body mass with a dual-energy x-ray absorptiometry (DXA) scan.

Subjects then initiate passive electrical muscle stimulation (EMS) delivered by a commercially available FDA approved neuromuscular stimulator ("EMPI 300PV" or its replacement, EMPI Continuum device obtained from EMPI, Inc., St Paul MN) 3 times a week to the quadriceps muscle groups (15 minutes on each side, 30 minutes total) while on hemodialysis. The duration of training will last for 4 months. Subjects will be monitored at regular intervals during the training to make sure they are doing the training correctly and they are not experiencing any problems.

At 2 and 4 months the subjects will undergo again have repeat assessment of the baseline testing as well as undergoing the standardized exercise stress test and a DXA scan.

At 4 months the subjects will all stop the passive exercise training and then will be followed up 1 month later to repeat assessment of all the baseline testing but will not undergoing the standardized exercise stress test and a DXA scan.

For subjects who agree the investigators will also perform a muscle biopsy under local anesthesia before and 4 hours after the first exercise training session and again at 2 and 4 months. This is used to measure messenger RNA response (gene expression testing) to tell what genes are activated during training.

The efficacy of the exercise training will be assessed by change in aerobic capacity measured by maximal oxygen consumption (peak VO2) and quadriceps muscle strength measured

The primary outcome measure will be whether exercise training improves measures of insulin resistance The investigators will also assess whether there is improvement in other inflammatory and oxidative stress cytokines in the blood stream and whether the training improved their physical performance or overall quality of life.

The total duration of the study for any patient is expected to be 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent
2. Currently on maintenance hemodialysis for end stage renal disease and expected to stay in the participating dialysis unit for at least 6 months.

Exclusion Criteria:

1. The presence of a cardiac pacemaker or presence of any other implanted electrical stimulation device
2. Uncontrolled hypertension as defined by a systolic BP >170 mmHg
3. Current presence of unstable angina
4. A heart attack (myocardial infarction) within the last month
5. Expected survival less than 6 months
6. Unsuitable for participation based on physician assessment
7. Pregnancy
8. Unwilling or unable to give informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07-29 (Actual); Primary Completion 2014-11-12 (Actual); Study Completion 2014-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley S Dixon, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from July 29, 2013 to March 25, 2014. All patients were from the outpatient dialysis program at the University of Iowa.
Pre-assignment Details: There was a 4 week care-optimization phase to make sure dialysis care was optimized before starting and to allow 2 separate measurements of baseline leg muscle strength. One patient withdrew from the study during this phase and did not complete the pre-EMS initiation measurements.
Period: Overall Study
Arm/Group | EMS Users in ESRD
Started | 7
Completed | 5
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- EMS Users: This was a longitudinal cohort study where all patients were entered into one study group receiving electrical muscle stimulation 3x/week for 30 minutes each session for a total of 16 weeks followed by a 4 week post-EMS study visit.
Arm/Group | EMS Users
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
History diabetes [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Muscle Strength Measured by a Belt-stabilized Portable Dynamometer
Description: Muscle strength was measured using a belt-stabilized hand held dynamometer (BSHHD) using a validated technique. Briefly, isometric knee extension strength (torque) was measured with patients seated on an elevated chair and their knees bent at about 90o of flexion (i.e., the legs hanging vertical). Patients are stabilized to the chair with straps around proximal thighs and waist. A dynamometer-stabilizing belt is passed around a bar secured behind the back legs of the chair and over a calibrated hand-held dynamometer that was placed against the anterior leg of the patient just proximal to the malleoli. The patient is asked to perform three leg extensions with the leg separated by 30 seconds of rest. The first effort is sub-maximal to get the patient accustom to the procedure. Then two full strength efforts are performed and used for calculation of average peak force (newtons, N) generated. The test is performed sequentially on both legs at each measurement session.
Time Frame: Baseline, Start EMS, 2 months and 4 months of EMS training, and 1 month post exercise
Population: Longitudinal prospective study of the effect of electrical muscle stimulation (EMS) on muscle strength.
Measure: Mean (Standard Deviation); unit: Force (Newtons)
Groups:
- Right Quadriceps Strength.: The effect of electrical muscle stimulation (EMS) on right quadriceps muscle strength will be assessed 5 times at baseline, pre-EMS training, at 8 and 16 weeks of EMS training and again 4 weeks after stopping EMS training. Right quadriceps muscle strength will be determined using a belt-stabilized portable dynamometer. This will determine if EMS produced an increase in right quadriceps strength after 8 and 16 weeks of training. It will also determine how rapidly the effect on muscle strength is lost after stopping EMS training.
- Left Quadriceps Strength: The effect of electrical muscle stimulation (EMS) on left quadriceps muscle strength will be assessed 5 times at baseline, pre-EMS training, at 8 and 16 weeks of EMS training and again 4 weeks after stopping EMS training. Left quadriceps muscle strength will be determined using a belt-stabilized portable dynamometer. This will determine if EMS produced an increase in left quadriceps strength after 8 and 16 weeks of training. It will also determine how rapidly the effect on muscle strength is lost after stopping EMS training.
Arm/Group | Right Quadriceps Strength. | Left Quadriceps Strength
Number analyzed (Participants) | 7 | 7
Force (Newtons)
  Baseline | 221.2 (81.8) | 227.4 (65.6)
  Start EMS: number analyzed (Participants) | 6 | 6
  Start EMS | 222.4 (80.4) | 213.5 (81.7)
  2 months EMS Training: number analyzed (Participants) | 6 | 6
  2 months EMS Training | 219.2 (73.6) | 213.9 (50.4)
  4 months EMS Training: number analyzed (Participants) | 6 | 6
  4 months EMS Training | 235.8 (59.9) | 204.7 (80.3)
  1 month Post-EMS training: number analyzed (Participants) | 6 | 6
  1 month Post-EMS training | 226.4 (63.8) | 151.9 (88.8)
Statistical Analysis 1: Comparison: Right Quadriceps Strength. vs Left Quadriceps Strength; Test type: Superiority; p = 0.999, Kruskal-Wallis — Threshold for statistical significance is P<0.05
Statistical Analysis 2: Comparison: Left Quadriceps Strength; Test type: Superiority; p = 0.768, Kruskal-Wallis

2. Secondary Outcome: Leg Composition by Dual Energy X-ray Absorptiometry (DXA).
Description: Advanced body composition analysis will be performed by DXA scan to measure regional fat and lean mass before starting EMS training and again after 2 and 4 months of EMS training. Specific areas of interest will be in determining whether EMS training produces the expected changes in thigh fat and muscle mass. The test is performed in the CRU at the University of Iowa using a Discovery A DXA scanner with the latest software version package (Hologic Inc., Bedford, MA). The advanced body composition analysis software package measures total regional body composition (cm2) using a validated technique that produces comparable results to a CT scan with less cost and radiation exposure.The total radiation dose is less than one tenth that of a standard CXR and equivalent to one-day exposure to natural background radiation. Patients will be asked to report to the CRU dressed metal-free (no zippers, jewelry, piercings, underwire bra, etc.). Each study will take approximately 30 minutes.
Time Frame: Baseline, 2 and 4 months of EMS training
Population: One of the 7 enrolled patients dropped out and did not undergo DXA measurements.
Measure: Mean (Standard Error); unit: cm squared
Groups:
- Right Total Thigh Mass: DXA measurement of total mass of right thigh
- Right Thigh Fat Mass: DXA measurement of fat mass of right thigh
- Right Thigh Lean Mass; Left Thigh Lean Mass: DXA measurement of lean mass of right thigh
- Left Total Thigh Mass: DXA measurement of total mass of left thigh
- Left Thigh Fat Mass: DXA measurement of fat mass of left thigh
Arm/Group | Right Total Thigh Mass | Right Thigh Fat Mass | Right Thigh Lean Mass | Left Total Thigh Mass | Left Thigh Fat Mass | Left Thigh Lean Mass
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
cm squared
  Baseline | 12458 (1501) | 4861 (1178) | 7369 (481) | 12492 (1498) | 4946 (1177) | 7301 (471)
  2 Months EMS Training | 12484 (1413) | 4835 (1042) | 7417 (542) | 12842 (1660) | 5109 (1164) | 7489 (607)
  4 Months EMS Training | 12540 (1553) | 4912 (1118) | 7392 (550) | 12831 (1706) | 5126 (1220) | 7453 (582)
Statistical Analysis 1: Comparison: Right Total Thigh Mass; Test type: Superiority; p = 0.869, Kruskal-Wallis
Statistical Analysis 2: Comparison: Right Thigh Fat Mass; Test type: Superiority; p = 0.813, Kruskal-Wallis
Statistical Analysis 3: Comparison: Right Thigh Lean Mass; Test type: Superiority; p = 0.978, Kruskal-Wallis
Statistical Analysis 4: Comparison: Left Total Thigh Mass; Test type: Superiority; p = 0.731, Kruskal-Wallis
Statistical Analysis 5: Comparison: Left Thigh Fat Mass; Test type: Superiority; p = 0.703, Kruskal-Wallis
Statistical Analysis 6: Comparison: Left Thigh Lean Mass; Test type: Superiority; p = 0.909, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 24 weeks on each patient. Adverse events were collected at the time of each study visit up to the last study visit which was 4 weeks after stopping the EMS training. Adverse events were also collected at any time we became aware of an adverse event during the period of the 24 weeks the patient was enrolled in the study.
Description: Questions asked of the participant at each visit: Is there a new medical diagnosis since the last visit? Specifically have you developed: Congestive heart failure (NYHA Grade); Myocardial infarction; Angina; Coronary angioplasty or bypass surgery; Carotid endarterectomy; Cardiac arrhythmias or conduction problems; Pericardial disease or pericarditis; Stroke or TIA; Claudication; Lower extremity angioplasty or bypass surgery; Amputation; Other new diagnosis; Any hospitalizations?
Groups:
- EMS Training Group: This is a longitudinal pilot study of electrical muscle stimulation (EMS training) on outcomes measures such as quadriceps strength. All participants under go the same protocol of EMS training. EMS is provided sequentially for 15 minutes to both the right and left quadriceps muscle groups three times a week while on hemodialysis. EMS is delivered to the quadriceps muscle groups using a neuromuscular electrical stimulator (using either the EMPI 300PV or its replacement, the Continuum device, EMPI, Inc). The device generates electrical impulses that are delivered to nerves stimulating the muscles through electrodes applied to the skin surface. Patients are taught how to place the adherent electrode pads over the quadriceps muscles on the upper thigh a few inches below the anterior iliac crest and just above the patella bilaterally. The patient will feel contraction of the muscles and may feel mild shortness of breath and tingling of the skin but otherwise is expected to tolerate the stimulation well. The first intervention will be observed through the entire treatment. If the patient feels excessively fatigued or other untoward signs the stimulator will be turned off until they feel better and then restarted to achieve the full treatment time.
Arm/Group | EMS Training Group
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EMS Training Group (N=7)
Transient ischemic attack (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03517553/Prot_SAP_000.pdf